CLINICAL TRIAL: NCT00622414
Title: A Phase I Study of VEGF Trap (NSC# 724770, IND# 100137) in Children With Refractory Solid Tumors
Brief Title: Aflibercept in Treating Young Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01062; NCI-2009-01062 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0714; CDR0000584050; NCI-08-C-0179; NCI-P08401; ADVL0714 (Other: COG Phase I Consortium); ADVL0714 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2008-02-22; First posted 2008-02-25 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — aflibercept

ARMS (1):
- Treatment (ziv-aflibercept) (Experimental): PART 1: Patients receive aflibercept IV over 1 hour on day 1. Treatment repeats every 14 days for 2 years in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive aflibercept until the maximum tolerated dose (MTD) is determined.
  PART 2: Patients receive aflibercept as in part 1 at 150% of the MTD determined in part 1. Treatment repeats every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept

INTERVENTIONS:
Biological: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap

SUMMARY:
This phase I trial is studying the side effects and best dose of aflibercept in treating young patients with relapsed or refractory solid tumors. Aflibercept may stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) or recommended phase II dose (RPTD) of aflibercept administered intravenously every 14 days in children with relapsed or refractory solid tumors.

II. To estimate the MTD or RPTD of aflibercept administered intravenously every 21 days in these patients.

III. To define and describe the toxicities of intravenous aflibercept administered on a 14-day and 21-day schedule, respectively.

IV. To characterize the pharmacokinetics of intravenous aflibercept in these patients.

SECONDARY OBJECTIVES:

I. To define, preliminarily, the antitumor activity of intravenous aflibercept within the confines of a phase I study.

OUTLINE: This is a multicenter study.

PART 1: Patients receive aflibercept IV over 1 hour on day 1. Treatment repeats every 14 days for 2 years in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive aflibercept until the maximum tolerated dose (MTD) is determined.

PART 2: Patients receive aflibercept as in part 1 at 150% of the MTD determined in part 1. Treatment repeats every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.

Blood samples are collected prior to treatment on day 1 of courses 1, 2, and 5 or 6 for pharmacokinetic studies.

After completion of study treatment, patients are followed for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy at original diagnosis or relapse (excluding intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of serum alpha-fetoprotein of beta-HCG)

  * Patients with recurrent or refractory solid tumors are eligible, including primary CNS tumors or patients with known CNS metastases
* Current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Measurable or evaluable disease
* No evidence of CNS hemorrhage on baseline MRI for patients with known CNS disease
* Karnofsky performance status (PS) 50-100% (for patients > 10 years of age) or Lansky PS 50-100% (for patients ≤ 10 years of age)

  * Neurologic deficits in patients with CNS tumors must have been relatively stable for a minimum of 1 week prior to study entry
  * Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients with solid tumors without bone marrow involvement must meet the following criteria:

  * ANC ≥ 1,000/mm³
  * Platelet count ≥ 100,000/mm³ (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
* Negative protein dipstick OR urine protein < 500 mg by 24-hour urine collection
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

  * 0.6 mg/dL for male and female patients 1 to < 2 years of age
  * 0.8 mg/dL for male and female patients 2 to < 6 years of age
  * 1.0 mg/dL for male and female patients 6 to < 10 years of age
  * 1.2 mg/dL for male and female patients 10 to < 13 years of age
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) for patients 13 to < 16 years of age
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) for patients ≥ 16 years of age
* Bilirubin ≤ 1.5 times upper limit of normal (U.N.) for age
* SEPT (ALT) ≤ 110 μ/L (approx. 2.5 times U.N.) (for the purpose of this study, the U.N. for SEPT is 45 μ/L)
* Serum albumin ≥ 2 g/dL
* PT/aPTT < 1.2 times U.N.
* Patients must have a diastolic blood pressure ≤ the 95th percentile for age and gender and not be receiving treatment for hypertension
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of active graft-vs-host disease
* No uncontrolled infection
* No serious or nonhealing wound, ulcer, or bone fracture
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to day 1 of study treatment
* No clinically significant cardiovascular disease within the past 6 months, including any of the following:

  * History of cerebrovascular accident
  * New York Heart Association class III-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Unstable angina pectoris
  * Pulmonary embolism
  * Deep vein thrombosis
  * Other thromboembolic events
* No evidence of a current bleeding diathesis or coagulopathy
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to other agents used in the study
* No significant traumatic injury within 4 weeks prior to day 1 of study treatment
* Must be able to comply with the safety monitoring requirements of the study in the opinion of the investigator
* Recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* No prior aflibercept
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea)
* At least 6 weeks since prior monoclonal antibodies
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 2 months since prior stem cell transplantation or rescue
* At least 3 months since prior total-body irradiation, craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 4 weeks since prior major surgical procedure, laparoscopic procedure, or open biopsy and no anticipation of need for major surgical procedures during the course of the study
* At least 48 hours since prior fine needle aspirate, central line placement, or subcutaneous port placement
* At least 1 week since prior core biopsy
* At least 1 week since prior and no concurrent hematopoietic growth factors
* At least 1 week since prior and no concurrent biologic agents
* At least 1 week since prior and no concurrent dexamethasone
* No concurrent antihypertensive medications for blood pressure control
* No concurrent anti-thrombotic or anti-platelet agents (e.g., warfarin [Coumadin ®],heparin, low molecular weight heparin, aspirin, and/or ibuprofen, or other NSAIDs)
* No concurrent medications known to inhibit platelet function or known to selectively inhibit cyclooxygenase-2 activity (e.g., all antipyretic and anti-inflammatory medications except acetaminophen)
* No other concurrent anticancer therapy, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy
* No other concurrent investigational drugs

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, defined as the maximum dose at which fewer than one-third of patients experience DLT during the initial 2 courses of therapy, graded according to NCI CTCAE version 3.0 | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Julie Park, Principal Investigator — COG Phase I Consortium
Locations (6):
- United States (6):
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington